CLINICAL TRIAL: NCT04906356
Title: Canadian Spontaneous Coronary Artery Dissection (SCAD) Study and Genetic Sub-study (Prospective, Observational Registry With 10 Year Follow-up)
Brief Title: Canadian SCAD Study
Status: Recruiting | Type: Observational
Sponsor: Cardiology Research UBC (Other)
Collaborators: John GB Mancini, MD (Unknown); Karin Humphries, DSc (Unknown)
Responsible Party: Principal Investigator, Jacqueline Saw, MD, Clinical Professor of Medicine, Cardiology Research UBC
Other Study IDs: H18-03039
Record Dates: First submitted 2021-04-16; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Spontaneous Coronary Artery Dissection; SCAD; Fibromuscular Dysplasia
Keywords: Fibromuscular displasia (FMD); Myocardial Infarction; Myocardial Infarction in women; Non-atherosclerotic coronary artery disease (NACAD); Myocardial Infarction with no obstructive coronary artery disease (MINOCA); SCAD; Spontaneous Coronary Artery Dissection
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous; Fibromuscular Dysplasia; Myocardial Infarction; MINOCA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva DNA sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Single group observational study
  Interventions: Genetic: Genetic sub-study

INTERVENTIONS:
Genetic: Genetic sub-study — One time saliva sample collection

SUMMARY:
Natural history multicenter, prospective, observational registry with 10-year follow-up

DETAILED DESCRIPTION:
Spontaneous coronary artery dissection (SCAD) is an under-diagnosed and poorly understood condition that frequently affects young women without conventional cardiovascular (CV) risk factors and can result in myocardial infarction (MI), cardiac arrest, and death. This condition has not been adequately studied, and there are no randomized controlled trials to guide treatment. Furthermore, SCAD has been frequently misdiagnosed due to the current "gold-standard" coronary angiography limitations. As such, there are uncertainties with the diagnosis and management of SCAD patients. Therefore, the investigators propose a large prospective multicenter Canadian SCAD Study to ascertain the natural history of predisposing arteriopathies and treatment strategy on short and long-term CV outcomes to design future randomized controlled trials.

This is a multicenter, prospective, international, observational natural history study with a planned total enrolment of 3,000 patients with SCAD. The investigators plan to recruit patients from major cardiac catheterization centers across Canada and several centers in the United States and internationally. The research team successfully enrolled 750 patients prospectively in the "Canadian SCAD Cohort Study" from 22 sites in North America. This current study will be an extension of that study, now named the "Canadian SCAD Study." It will continue enrolment for a total of 3,000 patients internationally (from >35 sites). Detailed baseline demographics, targeted history for precipitating stressors and predisposing conditions, and investigations for predisposing conditions will be performed during the study. Patients will be prospectively followed long-term for up to 10 years for CV events. The study is approved, allowing potential participants to be enrolled using an electronic consent form irrespective of their geographic location and directly communicating with the study team at UBC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted with ACS (STEMI, NSTEMI or unstable angina)
2. Documented SCAD on a coronary angiogram (including diagnosis with OCT or IVUS)

Exclusion Criteria:

1. Patients where SCAD is attributed to atherosclerotic coronary artery disease, with atherosclerotic coronary artery disease stenosis ≥50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with ACS (STEMI, NSTEMI or unstable angina) and diagnosed with SCAD during direct coronary angiography. The study imaging corelab will review all films before participant enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2033-12-01 (Estimated); Study Completion 2033-12-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital CV outcomes | From date of hospital admission to discharge up to 8 weeks
  Composite (Death, MI, CVA, Unplanned revascularization, Heart failure)
Long-term CV outcomes | at 10 Years post index event
  Composite (Death, MI, CVA, Revascularization, Heart failure)

SECONDARY OUTCOMES:
Arterial healing post SCAD | at 6 weeks post discharge post index event
  Angiographic healing
Coronary revascularization success | During index hospitalization
  Composite (TIMI 3 flow, <50% stenosis, and no residual dissection)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Saw, MD, Principal Investigator — Cardiology Research UBC / Vancouver General Hospital
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saw J, Starovoytov A, Humphries K, Sheth T, So D, Minhas K, Brass N, Lavoie A, Bishop H, Lavi S, Pearce C, Renner S, Madan M, Welsh RC, Lutchmedial S, Vijayaraghavan R, Aymong E, Har B, Ibrahim R, Gornik HL, Ganesh S, Buller C, Matteau A, Martucci G, Ko D, Mancini GBJ. Canadian spontaneous coronary artery dissection cohort study: in-hospital and 30-day outcomes. Eur Heart J. 2019 Apr 14;40(15):1188-1197. doi: 10.1093/eurheartj/ehz007. PMID 30698711